CLINICAL TRIAL: NCT01728246
Title: A Randomized Controlled Trial on the Efficacy, Safety and Quality of Life Effects of Add-on Tramadol/Paracetamol Combination in Chronic Osteoarthritis
Brief Title: An Efficacy, Safety and Effects on Quality of Life of Tramadol/Paracetamol as Add-on Therapy in Chronic Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013696; TRAMAPNAP4002
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Results first posted 2013-01-14 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Celecoxib; Tramadol; Paracetamol
MeSH Terms: conditions — Osteoarthritis | interventions — Tramadol; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tramadol/Paracetamol (APAP) (Experimental)
  Interventions: Drug: Tramadol/Paracetamol (APAP)
- Non-Tramadol/APAP (Active Comparator)
  Interventions: Drug: Non-Tramadol/APAP

INTERVENTIONS:
Drug: Tramadol/Paracetamol (APAP) — Celecoxib 200 milligram (mg) once daily for 4 weeks and fixed dose combination of Tramadol 37.5 mg/Paracetamol 325 mg thrice daily for 4 weeks as add-on therapy.
  Arms: Tramadol/Paracetamol (APAP)
Drug: Non-Tramadol/APAP — Celecoxib 200 mg alone once daily for 4 weeks.
  Arms: Non-Tramadol/APAP

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and effects on Quality of Life (QOL) of tramadol/paracetamol (APAP) as an add-on therapy (medication taken in addition to another medication) in Filipino participants with chronic (lasting a long time) osteoarthritis (disorder, which is seen mostly in older persons, in which the joints become painful and stiff).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (study drug assigned by chance), controlled study to evaluate the efficacy, safety and effects on QOL of tramadol/APAP as an add-on therapy in Filipino participants suffering from chronic pain because of chronic osteoarthritis. Participants will be randomly assigned to 2 groups: tramadol/APAP group and non tramadol/APAP group. Participants in tramadol/APAP group will receive celecoxib 200 milligram (mg) and fixed dose combination of tramadol (37.5 mg)/APAP (325 mg) as add on therapy, while the participants in non-tramadol/APAP group will receive celecoxib 200 mg only. The total duration of the study will be 4 weeks. The participants in both the groups will be given celecoxib 200 mg once daily for 4 weeks. In addition, the participants in the tramadol/APAP group will be given add-on tramadol/APAP doses 3 times a day for 4 weeks. Participants will be asked to return for follow-up at Weeks 2 and 4. Efficacy will be assessed using 100 millimeter (mm) Visual Analog Scale (VAS) while QOL will be assessed using the Oswestry Disability Index (ODI). Participant safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic osteoarthritis of knee or hip for greater than (>) or equal to (=) 1 year (based on the American College of Rheumatology (ACR) diagnostic criteria for osteoarthritis), who are experiencing at least moderate osteoarthritis pain (>=50 millimeter [mm] in 100 mm Visual Analog Scale [VAS])
* On any Cyclooxygenase - 2 (COX-2) inhibitors for at least 2 weeks preceding the study
* Women with childbearing potential must have negative pregnancy test
* Women of child bearing potential must agree to use accepted methods of contraception
* Participant has signed the written informed consent form

Exclusion Criteria:

* Participants taking Monoamine oxydase (MAO) inhibitors, neuroleptics or drugs for seizures
* Severe hepatic impairment (the impaired ability of the liver to fulfill its role in metabolism)
* On maintenance tramadol and/or paracetamol(APAP)
* On sedative hypnotics, short-acting analgesics, topical medications and anesthetics, and/or muscle relaxants
* Pregnant, lactating or breastfeeding participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical trial, Study Director — Janssen Pharmaceutica
Locations (1):
- Janssen Philippines, Paranaque City, National Capital Region, Philippines

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol/Paracetamol (APAP): Celecoxib 200 milligram (mg) administered orally once daily for 4 weeks and fixed dose combination of tramadol 37.5 mg/paracetamol 325 mg administered orally thrice daily for 4 weeks as add-on therapy.
- Non-Tramadol/APAP: Celecoxib 200 mg administered orally once daily for 4 weeks.
Period: Overall Study
Arm/Group | Tramadol/Paracetamol (APAP) | Non-Tramadol/APAP
Started | 242 | 231
Completed | 206 | 195
Not Completed | 36 | 36
Not completed — Participant needed rescue medication | 1 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 23 | 22
Not completed — Lack of Efficacy | 1 | 1
Not completed — Adverse Event | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol/Paracetamol (APAP) | Non-Tramadol/APAP | Total
Number analyzed (Participants) | 242 | 231 | 473
Age Continuous [Mean (Standard Deviation); unit: years] | 61.991 (12.084) | 62.40 (12.437) | 62.19 (12.248)
Sex/Gender, Customized [Number; unit: participants]
  Female | 171 | 177 | 348
  Male | 69 | 53 | 122
  Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Analogue Scale for Pain (VAS-pain) Score at Week 2
Description: VAS is a 100 millimeter (mm) scale. Intensity of pain range: 0 mm=no pain to 100 mm=worst possible pain. Change=scores at observation minus score at baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and Week 2
Population: Intent-to-treat (ITT) population included all the participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tramadol/Paracetamol (APAP) | Non-Tramadol/APAP
Number analyzed (Participants) | 242 | 231
mm
  Baseline | 71.86 (13.485) | 68.03 (13.77)
  Change at Week 2 | -29.721 (16.936) | -21.972 (12.906)
Statistical Analysis 1: Comparison: Tramadol/Paracetamol (APAP) vs Non-Tramadol/APAP; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Primary Outcome: Change From Baseline in VAS-pain Score at Week 4
Description: VAS is a 100 mm scale. Intensity of pain range: 0 mm=no pain to 100 mm=worst possible pain. Change=scores at observation minus score at Baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and Week 4 Last Observation Carried Forward (LOCF)
Population: ITT population included all the participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy assessment. LOCF method was used.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tramadol/Paracetamol (APAP) | Non-Tramadol/APAP
Number analyzed (Participants) | 242 | 231
mm | -45.027 (19.963) | -34.266 (15.665)
Statistical Analysis 1: Comparison: Tramadol/Paracetamol (APAP) vs Non-Tramadol/APAP; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

3. Primary Outcome: Change From Baseline in Oswestry Disability Index (ODI) Score at Week 2
Description: The ODI is a low back pain-specific, validated instrument that consists of questions related to limitations in performing specific activities of daily living and 1 question related to pain intensity. The ODI is a self-administered questionnaire that is usually completed in less than 5 minutes. The ODI consists of 10 sections. Each section consists of 6 statements ranked from 0 to 5 (0=good to 5=worse). A higher score represents greater disability.
Time Frame: Baseline and Week 2
Population: Data was not analyzed at Week 2 as time frame was too short to assess Quality of Life (QOL) by ODI score.
Arm/Group | Tramadol/Paracetamol (APAP) | Non-Tramadol/APAP
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change From Baseline in ODI Score at Week 4
Description: as for outcome 3
Time Frame: Baseline and Week 4 (LOCF)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol/Paracetamol (APAP) | Non-Tramadol/APAP
Number analyzed (Participants) | 242 | 231
units on a scale
  Baseline | 58.24 (17.034) | 57.23 (16.780)
  Change at Week 4 (LOCF) | -19.102 (15.103) | -15.177 (13.328)
Statistical Analysis 1: Comparison: Tramadol/Paracetamol (APAP) vs Non-Tramadol/APAP; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

5. Primary Outcome: Percentage of Participants Who Discontinued Because of Rescue Medication
Description: Rescue medications are medicines that may be administered to the participants when the efficacy of the study drug is not satisfactory, or the effect of the study drug is too great and is likely to cause a hazard to the participant, or to manage an emergency situation.
Time Frame: Baseline up to Week 4
Population: ITT population included all the participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Tramadol/Paracetamol (APAP) | Non-Tramadol/APAP
Number analyzed (Participants) | 242 | 231
percentage of participants | 0.41 | 2.16

6. Primary Outcome: Time to Discontinuation Because of Rescue Medication
Description: as for outcome 5
Time Frame: Baseline up to Week 4
Population: Time to discontinuation because of rescue medication was not analyzed, because dates when the rescue medication was given were not properly filled out in the forms, hence the exact time to discontinuation because of rescue medication could not be determined or analyzed.
Arm/Group | Tramadol/Paracetamol (APAP) | Non-Tramadol/APAP
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent until 30 days after the last dose of study medication
Arm/Group | Tramadol/Paracetamol (APAP) | Non-Tramadol/APAP
Serious Adverse Events (participants affected / at risk) | 1/242 | 1/231
Other Adverse Events (participants affected / at risk) | 19/242 | 10/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol/Paracetamol (APAP) (N=242) | Non-Tramadol/APAP (N=231)
Severe Hypertension (General disorders) | 1 | 0
Generalized Body Rashes (General disorders) | 1 | 0
Dizziness / Nausea (General disorders) | 1 | 0
Vaginal Bleeding (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol/Paracetamol (APAP) (N=242) | Non-Tramadol/APAP (N=231)
Drowsiness (General disorders) | 5 | 0
Abdominal Pain (General disorders) | 4 | 1
Dizziness / Nausea (General disorders) | 10 | 2
Vertigo (General disorders) | 0 | 2
Tachycardia (General disorders) | 0 | 1
Increase Pain (General disorders) | 1 | 0
Increase Swelling (General disorders) | 1 | 0
Dyspepsia (General disorders) | 0 | 1
Vomitting (General disorders) | 1 | 0
Palpitation (General disorders) | 0 | 1
Onset of Pain Contralateral to the Reference Point (General disorders) | 1 | 0
Leg Heaviness (General disorders) | 0 | 1
Headache (General disorders) | 0 | 1
Flatulence (General disorders) | 1 | 1
Cough (General disorders) | 0 | 1
Chest Tightening (General disorders) | 1 | 0
Sensation of Heat (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No